CLINICAL TRIAL: NCT06450483
Title: Comparing the Effects of Different Auricular Vagus Nerve Stimulation (AVNS) Parameters on Neck Pain Intensity, Heart Rate Variability (HRV), and Balance in Collegiate Athletes: A Randomized Comparative Effectiveness Design
Brief Title: Compare the Effects of Different AVNS Parameters on Neck Pain, HRV, Balance in Collegiate Atheletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Tamer Mohamed Shousha, Associate Professor, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AVNS on HRV and balance
Record Dates: First submitted 2024-05-27; First posted 2024-06-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Neck Pain; Heart Rate Variability; Balance
Keywords: AVNS; HRV; Balance; Neck Pain; Collegiate athletes
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Random allocation of two groups
Who Masked: Participant
Masking Description: the participants were masked in regards to the group they are in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular vagus stimulation in Group 1 (Experimental): Frequency: 25 Hz applied on the tragus of the ear, pulse length: 250 μs. A total of 4 sessions (2 sessions for 2 weeks). The sessions will be consistent with every participant where they were given their sessions on the same days every week.
  Interventions: Device: Auricular vagus nerve stimulation
- Auricular vagus stimulation in Group 2 (Experimental): Frequency: 10 Hz on the tragus of the ear, pulse length: 250 μs.A total of 4 sessions (2 sessions for 2 weeks). The sessions will be consistent with every participant where they will be given their sessions on the same days every week.
  Interventions: Device: Auricular vagus nerve stimulation

INTERVENTIONS:
Device: Auricular vagus nerve stimulation — Auricular vagal nerve stimulation using TPN dual channel TENS will be used for the study.The device used to stimulate is a conventional TENS. The stimulation is by applying a clip electrode placed on the tragus of the left ear and a second electrode applied on the left upper trapezius of the participant which will then stimulate the vagus nerve.Auricular vagus nerve stimulation session will be applied for 15 minutes. Participant is seated and relaxed.After the first session ended; heart rate will be measured and recorded once again to see the effect of the VNS.
  Before the last AVNS session started; heart rate will be measured and recorded. The participants' vagus nerve is then stimulated for 15 minutes.
  Other Names: TPN Dual Channel TENS

SUMMARY:
This study looks at how auricular vagus nerve stimulation (AVNS) affects neck pain, heart rate variability, and balance in college athletes, additionally, if different settings of auricular vagus nerve stimulation (AVNS) affect neck pain, heart rate variability, and balance in college athletes. The participants will be split into two groups, each receiving AVNS with different settings.

The study hypothesizes that vagus nerve stimulation (VNS) will reduce pain perception in college athletes. It is expected that auricular vagus nerve stimulation (AVNS) will decrease heart rate variability (HRV) in this population. Additionally, it is anticipated that college athletes undergoing AVNS will exhibit improved balance. The Investigators also believe that AVNS will decrease neck pain and enhance neck function. Finally, it is proposed that different AVNS parameters will have varying effects on pain intensity, HRV, and balance in collegiate athletes.

DETAILED DESCRIPTION:
This study investigated whether AVNS affects pain intensity, HRV, and balance in collegiate athletes with neck pain. Additionally, whether different AVNS parameters have different effects on pain intensity, HRV, and balance in collegiate athletes with neck pain? the objective of the study is to :

1. Investigate the effect of different AVNS parameters on pain intensity, HRV, and balance in collegiate athletes with neck pain.
2. Examine the effects of AVNS on heart rate variability in collegiate athletes.
3. Examine the effect of AVNS on balance in collegiate athletes.

The participants are assigned to two groups receiving distinct AVNS parameter sets. The study used five tools:

1. The International Physical Activity Questionnaire (IPAQ), 1998
2. Neck Pain Disability Index Questionnaire (Physio Therapy 1980)
3. Biodex Balance System SD (Biodex Medical Systems, Inc
4. Conventional TENS (TPN Dual Channel TENS)
5. Pulse Oximeter

Intervention Group 1: Participants in this category will undergo an auricular vagus nerve stimulation using the following parameters: Frequency: 25 Hz applied on the tragus of the ear, pulse length: 250 μs. Intervention Group 2: Participants in this category will undergo an auricular vagus nerve stimulation but with slightly different parameters: Frequency: 10 Hz on the tragus of the ear, pulse length: 250 μs. A total of 4 sessions (2 sessions for 2 weeks). The sessions will be consistent with every participant where they will be given their sessions on the same days every week.

The study hypothesizes that vagus nerve stimulation (VNS) will reduce pain perception in college athletes. It is expected that auricular vagus nerve stimulation (AVNS) will decrease heart rate variability (HRV) in this population. Additionally, it is anticipated that college athletes undergoing AVNS will exhibit improved balance. The researchers also believe that AVNS will decrease neck pain and enhance neck function. Finally, it is proposed that different AVNS parameters will have varying effects on pain intensity, HRV, and balance in collegiate athletes.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male and female Healthy collegiate athletes based in UAE
* Age range: 18-26 years
* Physical activity level: High score on the International Physical Activity Questionnaire
* BMI: Within the range of 20-25
* Neck pain level: Mild to moderate score on the Neck Pain Disability Index Questionnaire

Exclusion Criteria:

* Recent injury: Had an injury within the last three months
* Age: Over 26 years or below 18 years
* Physical activity level: Scored moderate or low on the International Physical Activity Questionnaire
* BMI: Above 25 or below 20
* Neck pain level: Scored severe on the Neck Pain Disability Index Questionnaire

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-07-03 (Estimated); Study Completion 2024-07-08 (Estimated)

PRIMARY OUTCOMES:
Neck pain | up to 6 weeks
  Numerical Pain Rating Scale( 0 no pain and 10 severe pain)
Neck pain disability | up to 6 weeks
  Neck pain disability Index (0-4:No Disability, 5-14:Mild Disability,15-24:Moderate Disability,25-34:Severe Disability, and above 34: Complete Disability)
Balance | up to 6 weeks
  Biodex Balance device to measure the dynamic balance test and limits of stability test
Heart Rate | up to 6 weeks
  Pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Tamer M Shousha, PhD, Principal Investigator — Associate professor
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates